CLINICAL TRIAL: NCT01740869
Title: Autologous Bone Marrow Stem Cells for Children With Autism Spectrum Disorders
Acronym: Autism
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hospital Universitario Dr. Jose E. Gonzalez (Other)
Responsible Party: Principal Investigator, M.D Laura Villarreal Martinez, Hematology Service, Hospital Universitario Dr. Jose E. Gonzalez
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: HE12-021; Autism uanl (Other: Autism uanl)
Record Dates: First submitted 2012-11-22; First posted 2012-12-04 (Estimated); Last update posted 2025-09-16 (Actual); Status verified 2025-03

CONDITIONS: Autism; Autism Spectrum
Keywords: autism; autism spectrum; stem cells; children
MeSH Terms: conditions — Autistic Disorder | interventions — Observation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | US Export: No

ARMS (2):
- Patients (Experimental): Children with autism spectrum disorder who will receive intrathecal infusion of autologous CD34+ hematopoietic stem cells after G-CSF stimulation and bone marrow harvest.
  Interventions: Biological: Autologous Intrathecal Hematopoietic Stem Cells
- Control (Other): Children with autism spectrum disorder who will be observed for 6 months and evaluated with CARS and IDEA scales, with option to crossover to the experimental arm afterwards.
  Interventions: Other: Observation with IDEA and CARS Scales

INTERVENTIONS:
Biological: Autologous Intrathecal Hematopoietic Stem Cells — Patients will be stimulated with granulocyte colony-stimulating factor (G-CSF) for 3 consecutive days. Bone marrow will be harvested, processed to isolate CD34+ hematopoietic stem cells and reduce red blood cells. An inoculum of 5-10 mL will then be infused intrathecally into the cerebrospinal fluid.
  Arms: Patients
Other: Observation with IDEA and CARS Scales — Participants will be observed for 6 months without active intervention. They will be evaluated using the Childhood Autism Rating Scale (CARS) and the IDEA scale at baseline, 30 days, and 180 days. After 6 months, participants may crossover to the experimental arm.
  Arms: Control

SUMMARY:
The purpose of this study is to determine whether the plasticity of autologous intrathecal hematopoietic cells would improve the neurologic and the social skills of pediatric patients with autism spectrum disorders.

DETAILED DESCRIPTION:
There is accumulating evidence that shows that the administration of hematopoietic cells into the brain in the patients with spectrum autism could help in the physiopathology of the illness.

It has been found that after introducing hematopoietic cells in the subarachnoid space of the spinal cord, these cells may be transported through the cerebrospinal fluid and can be delivered more efficiently to the injured area, when compared to the intravenous route.

Patients will be stimulated for 3 consecutive days with granulocyte colony stimulating factor (G-CSF) and then their bone marrow will be harvested according to their weight. Bone marrow will be processed in order to obtain CD34+ cells and minimize the amount of red blood cells. An inoculum of 5 to 10mL of stem cells will be infused intrathecally. Patients will be evaluated with two scales "CARS" and the "IDEA" also we will check the clinical history. On days 0, 30 and 180.

ELIGIBILITY:
Inclusion Criteria: Children aged 5 to 15 years, Diagnosis of Autism Spectrum Disorder (ASD) confirmed by DSM-5 criteria, Ability to comply with study procedures, including assessments with CARS and IDEA scales, Written informed consent obtained from parents or legal guardians.

Exclusion Criteria: Presence of severe neurological disorders other than ASD, History of immunodeficiency or hematologic disorders, Active infection at the time of enrollment, Previous treatment with intrathecal stem cells, Any medical condition that, in the investigator's judgment, would make participation unsafe.

Ages: 5 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Actual)
Dates: Start 2012-11 (Actual); Primary Completion 2016-11 (Actual); Study Completion 2017-10 (Actual)

PRIMARY OUTCOMES:
Change in Childhood Autism Rating Scale (CARS) score | Baseline, 30 days, and 180 days
  CARS scale will be used to evaluate changes in autistic behavior and social interaction after treatment. Participants will be assessed at baseline, 30 days, and 180 days to measure improvement following the intrathecal infusion of autologous CD34+ hematopoietic stem cells.

SECONDARY OUTCOMES:
Change in IDEA scale score | Baseline, 30 days, and 180 days
  IDEA scale will assess developmental and social abilities in participants. Measurements will be taken at baseline, 30 days, and 180 days to evaluate the effect of treatment on developmental progress.

CONTACTS AND LOCATIONS:
Locations (1):
- Hematology Service, Hospital Universitario Dr. Jose E. Gonzalez, Monterrey, Nuevo León, Mexico

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Siniscalco D, Sapone A, Cirillo A, Giordano C, Maione S, Antonucci N. Autism spectrum disorders: is mesenchymal stem cell personalized therapy the future? J Biomed Biotechnol. 2012;2012:480289. doi: 10.1155/2012/480289. Epub 2012 Feb 13. PMID 22496609
- [Background] Ichim TE, Solano F, Glenn E, Morales F, Smith L, Zabrecky G, Riordan NH. Stem cell therapy for autism. J Transl Med. 2007 Jun 27;5:30. doi: 10.1186/1479-5876-5-30. PMID 17597540
- [Background] Mehta T, Feroz A, Thakkar U, Vanikar A, Shah V, Trivedi H. Subarachnoid placement of stem cells in neurological disorders. Transplant Proc. 2008 May;40(4):1145-7. doi: 10.1016/j.transproceed.2008.03.026. PMID 18555135
- [Background] Hayashi T, Iwai M, Ikeda T, Jin G, Deguchi K, Nagotani S, Zhang H, Sehara Y, Nagano I, Shoji M, Ikenoue T, Abe K. Neural precursor cells division and migration in neonatal rat brain after ischemic/hypoxic injury. Brain Res. 2005 Mar 15;1038(1):41-9. doi: 10.1016/j.brainres.2004.12.048. PMID 15748871
- [Background] Nakatomi H, Kuriu T, Okabe S, Yamamoto S, Hatano O, Kawahara N, Tamura A, Kirino T, Nakafuku M. Regeneration of hippocampal pyramidal neurons after ischemic brain injury by recruitment of endogenous neural progenitors. Cell. 2002 Aug 23;110(4):429-41. doi: 10.1016/s0092-8674(02)00862-0. PMID 12202033
- [Background] Goldman SA, Schanz S, Windrem MS. Stem cell-based strategies for treating pediatric disorders of myelin. Hum Mol Genet. 2008 Apr 15;17(R1):R76-83. doi: 10.1093/hmg/ddn052. PMID 18632701
- [Background] Rempe DA, Kent TA. Using bone marrow stromal cells for treatment of stroke. Neurology. 2002 Aug 27;59(4):486-7. doi: 10.1212/wnl.59.4.486. No abstract available. PMID 12196638
- [Background] Felling RJ, Snyder MJ, Romanko MJ, Rothstein RP, Ziegler AN, Yang Z, Givogri MI, Bongarzone ER, Levison SW. Neural stem/progenitor cells participate in the regenerative response to perinatal hypoxia/ischemia. J Neurosci. 2006 Apr 19;26(16):4359-69. doi: 10.1523/JNEUROSCI.1898-05.2006. PMID 16624956
- [Background] Gordon PH, Yu Q, Qualls C, Winfield H, Dillon S, Greene PE, Fahn S, Breeze RE, Freed CR, Pullman SL. Reaction time and movement time after embryonic cell implantation in Parkinson disease. Arch Neurol. 2004 Jun;61(6):858-61. doi: 10.1001/archneur.61.6.858. PMID 15210522
- [Background] Kulbatski I, Mothe AJ, Nomura H, Tator CH. Endogenous and exogenous CNS derived stem/progenitor cell approaches for neurotrauma. Curr Drug Targets. 2005 Feb;6(1):111-26. doi: 10.2174/1389450053345037. PMID 15720218